CLINICAL TRIAL: NCT00198926
Title: Use of Modified Foods in the Dietary Treatment of Type II Diabetes Mellitus: Short Term Feeding Study
Brief Title: Type 2 Diabetes Controlled Eating Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: American Diabetes Association (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: ADA2000-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2001-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: covert v overt nutrition labeling
Behavioral: varying meal nutrition manipulation

SUMMARY:
A short-term feeding study in type 2 diabetics manipulating the fat and caloric values of meals to assess both compensation and glucose control, both covertly and overtly.

ELIGIBILITY:
Inclusion Criteria:

type 2 diabetic, age 18+, informed consent, able to eat 3 meals/day 1 day/week at clinic

Exclusion Criteria:

non-diabetic, type 1 diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2000-05; Study Completion 2001-08

PRIMARY OUTCOMES:
glucose control
caloric compensation

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States